CLINICAL TRIAL: NCT05531526
Title: A Phase 3 Double-blind, Randomized, Placebo-controlled, Multi-center Trial to Evaluate the Efficacy and Safety of AR1001 Over 52 Weeks in Participants With Early Alzheimer's Disease (Polaris-AD)
Brief Title: Phase 3, Double-blind, Randomized, Placebo-controlled Trial to Evaluate the Efficacy and Safety of AR1001 in Participants With Early Alzheimer's Disease (Polaris-AD)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AriBio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR1001-ADP3-US01
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: AR1001; AD; Early AD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A Phase 3 Double-blind, Randomized, Placebo-controlled, Multi-center Trial to Evaluate the Efficacy and Safety of AR1001 over 52 Weeks in Participants with Early Alzheimer's Disease
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind, randomized, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Active Comparator (Active Comparator): Active, AR1001 30 mg QD will be administered daily for 52 weeks during the Treatment Phase of the study. In the Extension Phase, all eligible participants who choose to participate will receive AR1001 30 mg QD for 52 weeks.
  Interventions: Drug: AR1001
- Group B - Placebo Comparator (Placebo Comparator): Placebo QD will be administered daily for 52 weeks during the Treatment Phase of the study. In the Extension Phase, all eligible participants who choose to participate will receive AR1001 30 mg QD for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR1001 — AR1001 Active Oral Tablet
  Arms: Group A - Active Comparator
Drug: Placebo — Placebo Oral Tablet
  Arms: Group B - Placebo Comparator

SUMMARY:
This AR1001-ADP3-US01 protocol is a double-blind, randomized, placebo-controlled, multi- center, parallel-group comparison pivotal Phase 3 study to evaluate the efficacy and safety of AR1001 for the treatment of participants with early AD.

DETAILED DESCRIPTION:
The purpose of this Study is to evaluate the efficacy and safety of AR1001 in participants with Early Alzheimer's Disease (AD).

AR1001 is a small molecule that has demonstrated its potential as a therapeutic agent for AD via its polypharmacological characteristics with multiple mechanisms to ameliorate AD pathology.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 55 to 90 years of age inclusive at the time of signing the informed consent form
2. Mild cognitive impairment or mild dementia consistent with AD defined by stages 3 to 4 according to the National Institute on Aging and Alzheimer's Association (NIA-AA) at Screening
3. Participants with a history of subjective cognitive and memory decline with onset within 5 years before Screening, confirmed by study partner.
4. Participants who have a MMSE score greater than or equal to 20
5. Participants with a CDR global rating of 0.5 or 1
6. Participants with a RBANS score based on the Delayed Memory Index (DMI) score less than or equal to 85
7. If an historic magnetic resonance imaging (MRI) is available, findings must exclude other causes of dementia.
8. Positive biomarker for brain amyloid pathology as indicated by assessment of at least one of the following:

   1. Current or historical CSF assessment with FDA-cleared assays, including Lumipulse® beta-amyloid ratio [1-42/1-40] ≤ 0.072, Elecsys® pTau 181/Aβ[1-42] greater than 0.023, Elecsys® tTau /Aβ[1-42] greater than 0.28, or other assays or cut-offs as they become FDA-cleared.
   2. Historical amyloid positron emission tomography (PET) assessment confirmed by the Sponsor or Designee.
9. Participants (or participant's legally authorized representative) and caregiver (s) who can sign an informed consent to participate in the study.
10. Participants who have one (or more) identified adult study partners (s) who, in the opinion of the Investigator, has sufficient contact with and knowledge about the participant as to be able to report knowledgably about the participant's cognition, function, behavior, and safety, and compliance with the protocol. The informant/care partner must be available by phone to provide information to the Investigator and study staff about the participant as well as agree to attend in-person clinic visits that require partner input for scale completion. The informant/care partner must be literate and provide informed consent and should be available for the duration of the study. The same informant/care partner is required to be consistent across all study visits except under rare, unavoidable circumstances (e.g., unexpected informant health crisis) that are approved by the Investigator and Sponsor.

Exclusion Criteria:

1. Participants who are female and are either pregnant, nursing, or of childbearing potential and not practicing effective contraception
2. Participants who have signs of significant delirium which, in the opinion of the Investigator, would interfere with this study
3. Participants who have any diagnosis of dementia or cognitive decline other than that related to AD, including, but not limited to concomitant history of significant head trauma, alcohol abuse, frontotemporal dementia, Huntington Disease, Parkinsonism (e.g., Parkinson's disease, Dementia with Lewy Bodies, etc.), significant cerebrovascular disease, and/or significant seizure disorder
4. Participants with any current psychiatric diagnosis if, in the judgment of the Investigator, the psychiatric disorder (e.g., schizophrenia) or symptom is likely to confound interpretation of drug effect, affect cognitive assessments, or affect the participant's ability to complete the study
5. Participants with a history of vascular dementia
6. Participants with evidence of other neurological conditions thought to interfere with the evaluations in this study
7. Participants with a history of myocardial infarction, unstable angina, coronary artery disease, and/or New York Heart Association (NYHA) class III or IV heart failure within the last 12 months
8. Participants with uncontrolled hypertension (systolic blood pressure (BP) >160 mmHg or diastolic BP > 95 mmHg) or hypotension (systolic BP <90 mmHg or diastolic BP <50 mmHg). Participants may undergo repeated testing to ensure that accurate BP readings are obtained
9. Participants with a body mass index (BMI) > 35 kg/m2
10. Participants with any of the following:

    1. elevation (>2.5x upper limit of normal [ULN]) of AST (aspartate aminotransferase, ALT (alanine transaminase, or total bilirubin (unless known prior history of Gilbert's syndrome)
    2. deficiency (< lower limit of normal [LLN]) of Vitamin B12
    3. known history of HIV (human immunodeficiency virus) positivity or positive test for HIV 1/2 at screening
    4. known history of Hepatitis C virus (HCV) or positive test for HCV antibody (HCVAb) at screening (unless negative on confirmatory PCR test)'
    5. positive test for Hepatitis B surface antigen (HBsAg)
    6. known history of neurosyphilis or positive test for RPR at screening
11. Participants who have history of cancer or malignant tumor within 5 years prior to screening with the exception of:

    1. Basal or squamous cell carcinoma of the skin or cervical dysplasia, which has been adequately treated
    2. In situ Grade 1 cervical cancer, fully treated at least 2 years prior to screening, and without recurrence.
    3. Prostate cancer, confined to the prostate gland, which has been adequately treated (e.g., surgery and/or radiation or watchful waiting) with normal or low and stable prostate-specific antigen (PSA) levels for 2 years prior to Screening
    4. Adequately treated non-metastatic breast cancer
12. Participants who in the opinion of the Investigator have an inadequately treated thyroid disorder
13. Participants with inherited degenerative retinal disease
14. Participants who have an undiagnosed or uncontrolled seizure disorder (and/or an epileptic syndrome), which has or could lead to cognitive impairment either from repeated seizures or the medications used to control the seizure disorder
15. Participants who are being treated, or likely to require treatment during the study, with any medications prohibited by the study protocol
16. Participants who have participated in any investigational drug or device trial within the previous 30 days or five half-lives of an investigational drug at Screening, whichever is longer
17. Participants taking an oral cholinesterase inhibitor and/or memantine not on a stable dose for at least 3 months prior to screening. Treatment and dosing should remain stable, with no changes throughout the trial.
18. Participants who have been and/or are currently being treated with anti-amyloid, anti-tau, or any other investigational therapies for AD
19. Participants who currently take any other PDE-5 Inhibitors (e.g., sildenafil)
20. Participants who are currently receiving (or unable to stop use for at least 14 days [2 weeks] prior to receiving the first dose of the AR1001 and throughout the study) prescription or nonprescription medications or other products known to be potent inhibitors of cytochrome P450 isozyme 3A4 (CYP3A4)
21. Alcohol or substance use disorder within the past 5 years according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
22. Participants who have previously participated in a clinical trial with AR1001
23. Participants, in the opinion of the Investigator, who are unsuitable to participate in the trial
24. Participants who in the opinion of the Investigator are at significant risk of suicide.
25. GDS-15 score greater than equal to 8 at Screening
26. Participants, in the opinion of the Investigator, who have any who have any contraindications to undergoing LP. Participants receiving ongoing anticoagulant therapy or antiplatelet therapy (other than aspirin and non-steroidal anti-inflammatory drugs [NSAIDs]) should also be excluded if it is considered unsafe to temporarily discontinue the therapy

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1535 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) | 52 weeks
  Change in the CDR-SB from Baseline to Week 52

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale, cognitive subscale (ADAS-Cog 13) | 52 weeks
  Change in ADAS-Cog 13 from Baseline to Week 52
Amsterdam-Instrumental Activities of Daily Living Questionnaire-Short Version (A-IADL-Q-SV) | 52 weeks
  Change in the A-IADL-Q-SV from Baseline to Week 52
Geriatric Depression Scale (GDS) | 52 weeks
  Change in the GDS from Baseline to Week 52
Mini-Mental Status Examination (MMSE) | 52 weeks
  Change in the MMSE from Baseline to Week 52

OTHER OUTCOMES:
Safety Analysis | 156 weeks
  * Frequency of treatment emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs)
  * Changes in C-SSRS (Columbia Suicide Severity Rating Scale)
Biomarker Analysis | 156 weeks
  Change in plasma/CSF biomarker levels from Baseline to Week 52 and the end of the Extension Phase.
Exploratory Analysis | 156 weeks
  Change in both primary and secondary endpoints from Baseline and Week 52 to the end of the extension study.

CONTACTS AND LOCATIONS:
Overall Officials: James Rock, Study Director — AriBio Co., Ltd.; Sharon Sha, MD, MS, Principal Investigator — Stanford University
Locations (198):
- United States (75):
  - IMA Clinical Research Phoenix, Phoenix, Arizona
  - Perseverance Research Center, LLC, Scottsdale, Arizona
  - Clinical Endpoints - N. Scottsdale, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Voyage Medical, Tempe, Arizona
  - Sutter Health's Palo Alto Medical Foundation, Burlingame, California
  - Neuro-Pain Medical Center, Fresno, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Esperanza Clinical, Murrieta, California
  - Valley Clinical Trials, INC, Northridge, California
  - Havana Research Institute, Pasadena, California
  - Kaizen Brain Center, San Diego, California
  - Adaptive Research, San Jose, California
  - The Neuron Clinic, San Marcos, California
  - Stanford Neuroscience Health Center, Stanford, California
  - Denver Neurological Research, Denver, Colorado
  - Mile High Research Center, Denver, Colorado
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Topaz Clinical Research, Apopka, Florida
  - BayCare Health System, Inc, Clearwater, Florida
  - Vertex Research Group, Clermont, Florida
  - Arrow Clinical Trial, Daytona Beach, Florida
  - Brainstorm Research - Loxahatchee, Loxahatchee Groves, Florida
  - ClinCloud LLC, Maitland, Florida
  - Verus Clinical Research, Corp, Miami, Florida
  - Vitae Research Center, LLC, Miami, Florida
  - Caro Medcenter and Community Research, Miami, Florida
  - Allied Biomedical Research Institute, Inc, Miami, Florida
  - Future Life Clinical Trials, Miami, Florida
  - Brainstorm Research, Miami, Florida
  - Meridian International Research, Inc, Miami Gardens, Florida
  - Charter Research - Orlando, Orlando, Florida
  - K2 Medical Research, Orlando, Florida
  - JEM Research Institute, Palm Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Angels Clinical Research Institute, Inc. - Tampa, Tampa, Florida
  - Charter Research - The Villages, The Villages, Florida
  - ClinCloud, LLC Melbourn, Viera, Florida
  - Conquest Research, Winter Park, Florida
  - iResearch -Atlanta, Atlanta, Georgia
  - Atlanta Neuroscience Institute, Atlanta, Georgia
  - Accel Research Sites, Decatur, Georgia
  - iResearch, Savannah, Georgia
  - Re:Cognition Health - Chicago, Chicago, Illinois
  - Tandem Clinical Research, New Orleans, Louisiana
  - BTC of New Bedford, New Bedford, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Headlands Research - Eastern MA, Plymouth, Massachusetts
  - Boston Paincare, Waltham, Massachusetts
  - Sharlin Health Neuroscience Research Center, Ozark, Missouri
  - Alivation, Lincoln, Nebraska
  - Wake Research- Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Dent Neuroscience Research Center, Amherst, New York
  - Mid-Hudson Medical Research, PLLC - New Windsor, New Windsor, New York
  - Triad Clinical Trials, Greensboro, North Carolina
  - AMC Research, LLC, Matthews, North Carolina
  - Accellacare of Winston-Salem, Triad Neurological Associates, Winston-Salem, North Carolina
  - NeuroScience Research Center, LLC, Canton, Ohio
  - American Clinical Research Institute, LLC, Dayton, Ohio
  - Rhode Island Mood and Memory REsearch, East Providence, Rhode Island
  - Health Concepts, Rapid City, South Dakota
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Center for Biomedical Research, LLC - Genesis Neuroscience Clinic, Knoxville, Tennessee
  - Gadolin Research LLC, Beaumont, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Cognition Health Corporation- Texas, Houston, Texas
  - Clinical Trial Network - Houston, Houston, Texas
  - Bhupesh Dihenia, MD, PA, Lubbock, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Cognition Health Corporation, Fairfax, Virginia
  - Integrated Neurology Services, Falls Church, Virginia
  - Kingfisher Cooperative, Spokane, Washington
  - Vaught Neurological Services, PLLC, Crab Orchard, West Virginia
  - Medical College of Wisconsin, Wauwatosa, Wisconsin
- Canada (10):
  - Centricity Research - Halifax, Halifax
  - Okanagan Clinical Trials, Kelowna
  - Parkwood Institute, London
  - Baycrest Academy for Research and Education, North York
  - Kawartha Centre - Redefining Healthy Aging, Peterborough
  - Centricity Research, Toronto
  - Sunnybrook Health Sciences Centre, Toronto
  - University Health Network-Toronto Western Hospital, Toronto
  - Royal Jubilee Hospital, Victoria
  - Medical Arts Health Research Group - West Vancouver, West Vancouver
- China (24):
  - Beijing Anding Hospital Capital Medical University, Beijing
  - Beijing Friendship Hospital,Capital Medical University, Beijing
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Sixth Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital of Central South University, Changsha
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Guangdong Provincial People's Hospital, Guangzhou
  - The Affiliated Brain Hospital Of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Anhui Provincial Hospital, Hefei
  - Tianjin Medical University General Hospital, Heping
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Huashan Hospital affiliated to Fudan University, Shanghai
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tongji Hospital Of Tongji University, Wuhan
  - Xuzhou Central Hospital, Xuzhou
- Czechia (8):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - NeuroHK s.r.o., Choceň
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Ambulance Smrkova ulice (A-Shine s.r.o.), Pilsen
  - FORBELI s.r.o, Prague
  - INEP Medical s.r.o., Prague
  - Neuropsychiatrie s.r.o., Prague
  - Vestra Clinics, Rychnov nad Kněžnou
- Denmark (3):
  - Sanos Clinic - Gandrup, Gandrup
  - Sanos Clinic - Herlev, Herlev
  - Sanos Clinic Syddanmark - Vejle, Vejle
- France (10):
  - CHU de Lille - Hopital Roger Salengro, Lille
  - AP-HM - Hopital de la Timone, Marseille
  - CHU de Nantes - Hopital Nord Laennec, Nantes
  - AP-HP Hopital Broca, Paris
  - AP-HP Hopital Lariboisiere, Paris
  - AP-HP Hopital Pitie-Salpetriere, Paris
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - CHRU de Strasbourg - Hopital de Hautepierre, Strasbourg
  - CHU de Toulouse - Hopital La Grave, Toulouse
  - HCL - Hopital des Charpennes, Villeurbanne
- Germany (6):
  - Universitaetsklinikum Aachen, AoeR, Aachen
  - Zentrum fuer klinische Forschung Dr. med. I. Schoell, Bad Homburg
  - Charite Universitaetsmedizin Berlin, Berlin
  - Bezirkskrankenhaus Guenzburg, Günzburg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Institut fuer Studien zur Psychischen Gesundheit (ISPG), Mannheim
- Italy (10):
  - Azienda Ospedaliero-Universitaria delle Marche, Ancona
  - IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
  - AOU Citta della Salute e della Scienza di Torino - Ospedale le Molinette, Torino
  - Pia Fondazione di Culto e Religione Cardinale Giovanni Panico, Tricase
- Netherlands (4):
  - Brain Research Center Den Bosch, 's-Hertogenbosch
  - Brain Research Center, Amsterdam
  - Amphia Ziekenhuis - Locatie Breda Molengracht, Breda
  - Brain Research Center Zwolle, Zwolle
- Poland (6):
  - KLIMED Marek Klimkiewicz, Bialystok
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Katowice
  - Osrodek Alzheimerowski Sp. z o.o, Ścinawa
  - ETG Neurosciences Sp. Z.o.o., Warsaw
  - NZOZ Wroclawskie Centrum Alzheimerowski, Wroclaw
- South Korea (24):
  - Seoul National University Bundang Hospital, Seongnam-si, Bundang-gu
  - Chonnam National University Hospital, Gwangju, Dong-Gu
  - Ewha Womans University Seoul Hospital, Seoul, Gangseo-gu
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Gachon University Gil Medical Center, Incheon, Namdong-Gu
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-gu
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul
  - Soonchunhyang University Hospital Cheonan, Cheonan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Hanyang University Guri Hospital, Guri-si
  - Uijeongbu St. Mary's Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Catholic Kwandong University International St.Mary's Hospital, Incheon
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St.Mary's Hospital, Seoul
  - Chung ang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Eunpyeong St.Mary's Hospital, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Ajou University Hospital, Suwon
- Spain (11):
  - Fundacio ACE - Institut Catala de Neurociencies Aplicades (Alzheimer Research Center Memory Clinic), Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Policlinica Gipuzkoa, San Sebastián
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (7):
  - Fulbourn Hospital, Cambridge
  - Cornwall Partnership NHS Foundation Trust, Cornwell
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Hammersmith Hospital, London
  - NeuroClin Glasgow, Motherwell
  - Warneford Hospital, Oxford
  - Southern Health NHS Foundation Trust, Southampton